CLINICAL TRIAL: NCT04174716
Title: An Open-label, Multi-center, Phase 1b/2a Basket Trial of IDX-1197 in Patients with Homologous Recombination Repair Mutated Solid Tumors
Brief Title: Basket Trial of IDX-1197, a PARP Inhibitor, in Patients with HRR Mutated Solid Tumors (VASTUS)
Acronym: VASTUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Idience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-VDP-102
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumors; Homologous Recombination Repair Gene Mutation; Homologous Recombination Deficiency
Keywords: HRR; 1197; venadaparib; IDX-1197

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IDX-1197 (Experimental): Patient will be receive IDX-1197HCl once daily for 28 continuous days
  Interventions: Drug: IDX-1197

INTERVENTIONS:
Drug: IDX-1197 — Until progression or unacceptable toxicity develops

SUMMARY:
This study is a Phase 1b/2a basket trial to assess safety and efficacy of IDX-1197 in patients with HRR mutation.

There are two parts to this study: Phase 1b, IDX-1197 dose-selection study to determine RP2D and Phase 2a, non-randomized parallel dose expansion study to confirm RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancers that have HRR mutation and are failed to standard therapy or for which standard or curative therapy does not exist or is not considered appropriate by the Investigator.
* Measurable disease according to RECIST, v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* Must have recovered from all side effects of their most recent systemic or local treatment (<CTCAE grade 3)
* Life expectancy greater than 12weeks

Exclusion Criteria:

* Prior treatment with PARP inhibitors
* Symptomatic CNS metastases
* History of or known carcinomatous meningitis
* Concurrent administration of any anti-cancer therapies other than those administered in this study
* Pregnant or lactating women
* Refractory nausea and vomiting, malabsorption, total gastrectomy, external biliary shunt or significant bowel resection that would preclude adequate absorption.
* Uncontrolled medical illness (such as infection requiring treatment with intravenous antibiotics)
* Severe or unstable angina, myocardial infarction or ischemia requiring coronary artery bypass graft or stent within the previous 6 months, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to enrollment or New York Heart Association (NYHA) Class II to IV heart disease.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
* Known hypersensitivity to IDX-1197 or any of the excipients of the product

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | Up to 24 weeks
  Confirmed objective response rate (ORR) determined by the Investigator using Response Evaluation Criteria In Solid Tumors, Version 1.1 (RECIST, v1.1).

CONTACTS AND LOCATIONS:
Locations (19):
- South Korea (19):
  - National Cancer Centre, Goyang, Gyeongggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Inje University Haeundae Hospital, Busan
  - Dong-a University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Cha University Bundang Medical Center, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided